CLINICAL TRIAL: NCT00005184
Title: Immunogenetic Factors of Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1062; R01HL033959 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypertension; Obesity; Diabetes Mellitus; Hypothyroidism
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypertension; Obesity; Diabetes Mellitus; Hypothyroidism

SUMMARY:
To assess the association of immunogenetic factors with onset of coronary heart disease and the interrelationship of these factors with standard coronary heart disease risk factors.

DETAILED DESCRIPTION:
BACKGROUND:

Although the familial clustering of coronary heart disease has been well documented, it is unclear as to whether the familial clustering can be explained by shared environmental factors by members of a family or by clustering of risk factors having a genetic component such as blood pressure, familial hyperlipidemia and/or diabetes. Studies indicate that a family history of coronary disease may be an independent risk factor. Major histocompatibility complex genetic markers to identify individuals at risk within a family may be useful. In 1985 when the study began, there was a paucity of data dealing with the interrelationship of family history, genetic markers, immunological markers, and traditional risk factors.

DESIGN NARRATIVE:

In this case-control study, the study population consisted of incident cases who presented to the Georgia Heart Clinic in La Grange, Georgia with coronary heart disease. The majority of the subjects were from three counties in mideastern Alabama and from counties in midwestern Georgia. All subjects had undergone diagnostic coronary angiography. A determination was made in patients and controls of the association of major histocompatibility complex genetic markers HLA-A, -B, -C, -DR, C4 and BF, C3, the restriction fragment length polymorphisms (RFLP's) flanking the apolipoprotein AI and insulin genes, presence of autoantibodies, and family history of coronary disease, diabetes, or hypothyroidism. The frequency of these variables was compared with the standard coronary risk factors of family history, hypertension, lipid abnormalities, lifestyle, Type A behavior, obesity and with diseases such as diabetes and hypothyroidism. An analysis was made of the strength of these variables for predicting those individuals at risk and whether there were variables which predict severity of disease based on 1, 2, or 3 vessel involvement.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-12; Study Completion 1989-11 (Actual)

REFERENCES:
- [Background] Go R, Acton R, Roseman J, Barger B, Perkins L, Vanichanan T, Moore P, Brand J, Gore T, Brennan J, Cousins L, Copeland R: Immunogenetic Risk Factors for Premature Coronary Artery Disease in Southeastern USA Population. Genome, 30:34, 1988
- [Background] Acton R, Bamberg R, Go R, Roseman J: Utilization of Genetic and Other Laboratory Test Results to Predict and Reduce the Risk of Disease. In: Proceedings of the Society of Prospective Medicine, 1988. 1988.
- [Background] Bamberg R, Copeland R, Barger B, Roseman J, Go R, Vanichanan C, Brand J, Moore P, Acton R: Genetic Risk Information as an Impetus to Health Related Behavioral Change. In: Proceedings of the Society of Prospective Medicine, 1988. 1988.
- [Background] Pancharuniti N, Lewis CA, Sauberlich HE, Perkins LL, Go RC, Alvarez JO, Macaluso M, Acton RT, Copeland RB, Cousins AL, et al. Plasma homocyst(e)ine, folate, and vitamin B-12 concentrations and risk for early-onset coronary artery disease. Am J Clin Nutr. 1994 Apr;59(4):940-8. doi: 10.1093/ajcn/59.4.940. PMID 8147342